CLINICAL TRIAL: NCT02283021
Title: Expression and Sequence of Calcium Channels in Non-small Cell Lung Carcinoma (NSCLC)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: CALCIUM-HMO-CTIL
Record Dates: First submitted 2014-10-05; First posted 2014-11-05 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: NSCLC
Keywords: expression of L-type calcium subunits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lung specimen biospsies are routinely taken from NSCLC patients and sent to pathological evaluation. We will obtain small samples from these biopsies from the pathologist, which are normally discarded. mRNA will be extracted from these samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NSCLC Patients: Sample biopsies from normal and cancerous lung tissue.
  Interventions: Other: A biopsy sample
- Patients without NSCLC: Sample biopsies from normal lung tissue.Control group.
  Interventions: Other: A biopsy sample

INTERVENTIONS:
Other: A biopsy sample — Sample tissue will be obtained from the routine biopsy taken for pathological evaluation. A pathologist will determine which part of the tissue will be forwarded for this study, to avoid any interference with the pathological evaluation.

SUMMARY:
Calcium is an extremely important ion used in our body for many processes. One of its tasks is to control gene expression. Cells intake calcium from their surroundings though special calcium channels located on the surface membranes of the cells.

The great many studies on such calcium channels were performed on excitable cells such as muscle, heart or neuronal cells, where the calcium ions are controlled by voltage. Surprisingly, not much is known about the identity of calcium subunits in non-excitable cells like epithelial cells (which compose most of the connective tissue in the body), liver cells, lung cells, immune system cells, etc.

Recently, the investigators have shown that calcium channels from muscles are, in fact, expressed in T cells of the immune system, where they are used for proliferation. The investigators postulated that probably other cell types, especially cancerous cell types, might be using these subunits similarly.

The aim of this study is to determine the identity and sequence of calcium subunits expressed in non-small cell Lung Carcinoma (NSCLC), which accounts for 80% of the worldwide lung cancer deaths.

DETAILED DESCRIPTION:
Initial examination of NSCLC cell lines determined that they express the mRNA of voltage gated calcium subunits, found normally in neurons. Furthermore sequence analysis of these subunits has shown that modifications have occurred.

The aim of the study in NSCLC patients is to sequence and clone the calcium channel subunits expressed in their tumor. Expression and Sequence will be compared between the normal and cancerous lung tissue for each patient.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC patients
* Patients without NSCLC
* Men or woman between 18-80 years of age

Exclusion Criteria:

* Pregnant woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with NSCLC and patients not diagnosed with NSCLC
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
mRNA expression and sequence of calcium channel subunits in NSCLC | up to 1 month per patient
  mRNA will be extracted from each sample biopsy followed by real time PCR analysis. If any calcium subunit is detected, semi quantitative PCR will be performed, PCR bands will be cloned and sequenced.

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Lamberg, PhD, Study Director — Hadassah Medical Organization